CLINICAL TRIAL: NCT01452061
Title: Understanding Genetic Differences Associated With Autism Spectrum and Attention Deficit/Hyperactivity Disorder
Brief Title: Evaluating the Validity of a Genetic Risk Assessment Tool in Identifying Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Thomas W. Frazier, Ph.D (Other)
Collaborators: IntegraGen SA (Industry)
Responsible Party: Sponsor-Investigator, Thomas W. Frazier, Ph.D, Center for Autism Research Director, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: CCF 11-949
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Autism Spectrum Disorder; Attention Deficit/Hyperactivity Disorder; Developmental Delay
Keywords: Autism Spectrum Disorder; Attention Deficit/Hyperactivity Disorder; Developmental Delay
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genetic material via a cheek swab will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ASD: Participants with autism spectrum disorder.
- ADHD/DD: Participants with attention deficit/hyperactivity disorder, developmental delay or psychiatric disorder.
- Siblings: Siblings without a developmental or psychiatric disorder.
- Control: Unrelated individuals without a developmental or psychiatric disorder.

SUMMARY:
There are three purposes to this study. The first purpose is to evaluate the value of a genetic test in determining risk for autism spectrum disorder. Processing for genetic samples will be completed at the Cleveland Clinic using research equipment provided by IntegraGen. The second purpose is to identify genetic changes that may be associated with autism spectrum disorder or attention deficit/hyperactivity disorder. The third purpose is to examine whether genetic differences and changes may predict which individuals benefit from medicine used to treat attention problems or other psychiatric difficulties.

Between 600-800 people are expected to participate in this study - approximately 300 individuals with an autism spectrum disorder, 75 individuals with attention deficit/hyperactivity disorder or another developmental or psychiatric disorder, 100 healthy siblings, and 125 unrelated individuals without a developmental or psychiatric disorder.

Study procedures will vary based upon the specific group participants are suspected to fall into (autism, attention deficit/hyperactivity disorder, psychiatric concerns/developmental delay, healthy sibling, or unrelated healthy control).

* All individuals will be asked to participate in a cheek swab (gently swabbing the inside of your cheek) to obtain cells used for genetic testing. Genetic material will be stored with identifiers such as numbers, letters or codes.
* Parents or caregivers will be asked to complete questionnaires that examine medical and family history as well as current symptoms and quality of life for the participant.
* Participants may undergo speech and language testing. This involves answering questions, looking at pictures or identifying items.
* Information recorded in participant medical records will be reviewed and collected for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autistic Disorder, Pervasive Developmental Disorder, or Asperger's Disorder or have a clinical diagnosis of another developmental or psychiatric disorder (developmental/psychiatric controls), or have no specific developmental or psychiatric diagnosis (healthy controls).
* Age 1 to 12.

Exclusion Criteria:

* For individuals with ASD and developmental concern controls, presence of a known or strongly suspected genetic disorder based on all available clinical data.
* Age less than 1 or greater than 12.
* Individuals for whom DNA is not available for analysis.
* Individuals for whom it is anticipated that they will not be available for follow-up at the Cleveland Clinic during the study period.
* Any medical diagnoses that might preclude participation in a low risk, non-interventional research study and any participant who at the discretion of the clinical investigator is not medically able to participate in the study (e.g., unable to comply with cheek swab or other procedure or has serious medical condition which precludes participation).

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: About 600 people will take part in this study - 300 individuals with an autism spectrum disorder, 75 individuals with attention deficit/hyperactivity disorder or another developmental or psychiatric disorder, 100 healthy siblings, and 125 unrelated individuals without a developmental or psychiatric disorder.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Autism Spectrum Disorder clinical diagnosis | March 2014

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Frazier, Ph.D., Principal Investigator — The Cleveland Clinic; Charis Eng, M.D., Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Autism, Cleveland, Ohio, United States

REFERENCES:
- See also: Cleveland Clinic Center for Autism Research Website — http://clevelandclinic.org/autismresearch